CLINICAL TRIAL: NCT01912573
Title: Nasal Naloxone for Narcotic Overdose
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Judith Feinberg (Other)
Responsible Party: Sponsor-Investigator, Judith Feinberg, Assoc Chair of Medicine, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N3OD; Ohio Division of EMS Board (Other Grant/Funding Number: Ohio Department of Public Safety)
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Drug Overdose
Keywords: heroin; prescription pain killers; narcotics
MeSH Terms: conditions — Drug Overdose | interventions — Naloxone; Injections, Intramuscular; Jupiter

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intranasal (IN) naloxone (Experimental): Intranasal (IN) naloxone as initial response to suspected opioid overdose
  Interventions: Drug: Intranasal (IN) naloxone
- Standard of Care (TAU) (Active Comparator): Standard of care (intravenous [IV], intramuscular [IM] or intraosseus [IO]delivery of naloxone) as initial response to suspected opioid overdose.
  Interventions: Drug: Intravenous (IV) naloxone; Drug: Intramuscular (IM) naloxone; Drug: Intraosseus (IO) naloxone

INTERVENTIONS:
Drug: Intranasal (IN) naloxone
  Other Names: Narcan
  Arms: Intranasal (IN) naloxone
Drug: Intravenous (IV) naloxone
  Other Names: Narcan
  Arms: Standard of Care (TAU)
Drug: Intramuscular (IM) naloxone
  Other Names: Narcan
  Arms: Standard of Care (TAU)
Drug: Intraosseus (IO) naloxone
  Other Names: Narcan
  Arms: Standard of Care (TAU)

SUMMARY:
The goal of this study is to determine if nasal naloxone is inferior to standard care for naloxone administration in a pre-hospital setting. Ambulance squads in Adams, Clermont, and Scioto counties in southern Ohio will be randomized to provide either standard care or nasal (IN) naloxone as the initial response to a suspected opioid overdose. Standard care includes administration of naloxone by intravenous (IV), intramuscular (IM) or intraosseus (IO) methods.

DETAILED DESCRIPTION:
This is a randomized, prospective trial that will compare clinical outcomes for parenteral naloxone according to the standard of care (TAU; administration via intravenous [IV], intramuscular [IM] or intraosseus [IO] delivery) versus intranasal [IN] for the prehospital emergency treatment of suspected opioid overdose. Ambulance squads in Adams, Clermont, and Scioto counties in southern Ohio will be randomized to administer either standard care or IN naloxone as the initial response to a suspected opioid overdose.

ELIGIBILITY:
Inclusion Criteria:

* Presence of hyperventilation or respiratory arrest OR
* EMS assessment that the person needs naloxone for possible opioid or unknown drug overdose

Exclusion Criteria:

* EMS assessment that the participant is less than 12 years old

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with adequate respiration within 10 minutes | 10 minutes after intervention administration

SECONDARY OUTCOMES:
Number of patients requiring second dose of naloxone | within 10 minutes of initial dose
Time to first naloxone administration | at baseline
  Time between emergency call and administration of naloxone.
Opioid Withdrawal Symptoms | baseline
Naloxone Adverse Events | 3 hours
Proportion of Patients breathing unassisted upon arrival to the hospital | within 1 hour
Days of hospitalization following naloxone administration | 7 days
Mortality rate | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Judith Feinberg, MD, Principal Investigator — University of Cincinnati
Locations (3):
- United States (3):
  - Clermont County, Batavia, Ohio
  - Scioto County, Portsmouth, Ohio
  - Adams County, West Union, Ohio